CLINICAL TRIAL: NCT05398263
Title: A Randomised, Double-Blind, Parallel-Group, Placebo-Controlled 28-week Phase 3 Efficacy and Safety Study of Tezepelumab in Reducing Oral Corticosteroid Use in Adults With Oral Corticosteroid Dependent Asthma (SUNRISE)
Brief Title: Tezepelumab Efficacy and Safety in Reducing Oral Corticosteroid Use in Adults With Oral Corticosteroid Dependent Asthma
Acronym: SUNRISE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was discontinued due to slow recruitment, resulting from evolving clinical practices that reduced the use of maintenance oral corticosteroids for severe asthma treatment. The termination decision was not related to safety concerns.
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5180C00024; 05398263 (Registry Identifier: ClinicalTrials.gov); 2023-504648-33 (Other: EU CT Number); 2023-504648-33-00 (Registry Identifier: CTIS); 2021-006691-17 (EudraCT Number)
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Asthma
Keywords: Asthma; Severe Asthma; Oral Corticosteroid Dependent Asthma; Tezepelumab; Phase 3 Study; Reducing Oral Corticosteroid
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 2:1 ratio to either tezepelumab or matching placebo both administered subcutaneously.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tezepelumab (Experimental): Tezepelumab subcutaneous injection, in an accessorised pre-filled syringe.
  Interventions: Biological: Tezepelumab
- Placebo (Placebo Comparator): Placebo subcutaneous injection, in an accessorised pre-filled syringe.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab subcutaneous injection
  Arms: Tezepelumab
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
A Randomised, Double-Blind, Parallel-Group, Placebo-Controlled 28-week Phase 3 Efficacy and Safety Study of Tezepelumab in Reducing Oral Corticosteroid Use in Adults with Oral Corticosteroid Dependent Asthma

DETAILED DESCRIPTION:
This is a multicentre, randomised, double-blind, placebo controlled, parallel group study designed to evaluate the efficacy and safety of tezepelumab in reducing oral corticosteroid use in adults with oral corticosteroid dependent asthma treated with maintenance OCS in combination with high dose inhaled corticosteroids (ICS) and long-acting β2 agonists (LABA), with or without other asthma controller therapies. Approximately 207 subjects will be randomized globally. Subjects will receive tezepelumab, or placebo, administered via subcutaneous injection using the accessorized pre-filled syringe (APFS), over a 28-week treatment period. The study also includes a post-treatment follow-up period of 12 weeks.

ELIGIBILITY:
Main inclusion criteria:

1. Participant must be 18 to 80 years of age.
2. Documented physician-diagnosed asthma for at least 12 months prior to Visit 1.
3. Participants must have received a physician-prescribed medium- or high-dose ICS for at least 12 months prior to Visit 1.
4. Participants must have received physician prescribed LABA and high dose ICS for at least 3 months prior to Visit 1.
5. Additional maintenance asthma controller medications are allowed. The use of these medications must be documented for at least 3 months prior to Visit 1.
6. Participants must have received OCS for the treatment of asthma for at least 6 months prior to Visit 1 and on a stable dose of between ≥7.5 to ≤ 30 mg (prednisone or prednisolone) daily or daily equivalent for at least 1 month prior to Visit 1.
7. Morning pre- bronchodilator (BD) FEV1 must be < 80% predicted normal at Visit 1 or Visit 2.
8. Evidence of asthma as documented by either:

   a)Post-BD responsiveness test result: FEV1 ≥12% and ≥200 mL documented either in the previous 60 months prior to or at Visit 1 or at Visit 2 or at Visit 3; OR b)Airway hyperresponsiveness (methacholine: provocative concentration that causes a positive reaction [PC20] of <8 mg/mL) documented in the 60 months prior to Visit 1.
9. Blood eosinophils at Visit 1 ≥150 cells/μL or documented EOS ≥300 cells/μL within 12 months prior to Visit 1.
10. Participants must have a history of at least 1 asthma exacerbation event within 24 months prior to Visit 1.
11. Participants must have received the optimised OCS dose for at least 2 weeks prior to randomisation.

Other inclusion criteria per protocol apply.

Main exclusion criteria

1. Any clinically important pulmonary disease other than asthma.
2. Any disorder that is not stable in the opinion of the Investigator and could: a. Affect the safety of the participant throughout the study; b. Influence the findings of the study or the interpretation; c. Impede the participant's ability to complete the entire duration of study.
3. History of cancer: a. Participants who have had basal cell carcinoma, localised squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible to participate in the study provided that curative therapy was completed at least 12 months prior to Visit 1; b. Participants who have had other malignancies are eligible provided that curative therapy was completed at least 5 years prior to Visit 1.
4. Asthma exacerbation, requiring use of systemic corticosteroids or increase in the maintenance dose of OCS finalized within 30 days prior to Visit 1.
5. Clinically significant infection requiring treatment with systemic antibiotics or antiviral medications finalized < 2 weeks before Visit 1 or during the run-in period.
6. Participants with evidence of active COVID-19 infection during run-in period and optimisation.
7. A helminth infection diagnosed within 6 months prior to Visit 1 that has not been treated with, or has failed to respond to, standard of care therapy.
8. A participant who is on SABA maintenance treatment within 30 days prior to Visit 1.
9. Current smokers or participants with smoking history ≥ 10 pack-years and participants using vaping products, including electronic cigarettes. Former smokers with a smoking history of <10 pack years and users of vaping or e-cigarette products must have stopped for at least 6 months prior to Visit 1 to be eligible.
10. Receipt of any marketed or investigational biologic agent within 4 months or 5 half-lives (whichever is longer) prior to Visit 1 or receipt of any investigational non-biologic agent within 30 days or 5 half-lives (whichever is longer) prior to Visit 1.
11. COVID-19 vaccination within 28 days prior to randomisation.
12. Tuberculosis requiring treatment within the 12 months prior to Visit 1.
13. During the optimisation period, asthma control reached at an OCS dose of <7.5 mg or >30 mg and/or 3 consecutive dose reductions after which asthma control was still obtained.

Other exclusion criteria per protocol apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Categorised percent reduction from baseline in the daily maintenance OCS dose at Week 28 whilst maintaining asthma control. | Baseline to Week 28
  Categorised percent reduction from baseline at Week 28. Percent change from baseline is defined as {final dose-baseline dose)/baseline dose}*100%, and the categories of percent change from baseline in daily OCS dose are defined as: ≥90% to ≤100% reduction, ≥75% to <90% reduction, ≥50% to <75% reduction, >0% to <50% reduction, and, no change or any increase.

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator (pre-BD) forced expiratory volume in 1 second (FEV1) at Week 28 | Baseline to Week 28
  Change from baseline in pre-BD FEV1 at Week 28. FEV1 is defined as the volume of air exhaled from the lungs in the first second of a forced expiration.
Proportion of subjects with 100% reduction from baseline in daily OCS dose at Week 28 | Baseline to Week 28
  Proportion of subjects with 100% reduction from baseline in daily OCS dose at Week 28. Percent change from baseline is defined as {(final dose-baseline dose)/baseline dose}*100%.
Proportion of subjects with daily OCS dose ≤5 mg at Week 28 | Week 28
  Proportion of subjects with daily OCS dose ≤5 mg at Week 28.
Proportion of subjects with ≥50% reduction from baseline in daily OCS dose at Week 28 | Baseline to Week 28
  Proportion of subjects with ≥50% reduction from baseline in daily OCS dose at Week 28. Percent change from baseline is defined as {(final dose-baseline dose)/baseline dose}*100%.
Annualised asthma exacerbation rate (AAER) over 28 weeks | Baseline to Week 28
  The annualized exacerbation rate is based on exacerbations reported by the investigator in the eCRF over 28 weeks.
Time to first asthma exacerbation | Baseline to Week 28
  Time to first asthma exacerbation.
Change from baseline in Asthma Control Questionnaire 6 (ACQ-6) score at Week 28 | Baseline to Week 28
  Change from baseline in ACQ-6 as compared to placebo at Week 28. The ACQ-6 captures asthma symptoms and short-acting β2-agonist use via subject-report. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The ACQ-6 score is the mean of the responses.
Change from baseline in weekly mean home peak expiratory flow (PEF) (morning and evening) at Week 28 | Baseline to Week 28
  Change from baseline in weekly mean morning and evening peak expiratory flow (PEF) as compared to placebo at Week 28. Home PEF testing will be performed by the subject in the morning upon awakening and in the evening at bedtime using an electronic, hand-held spirometer. Each timepoint is calculated as weekly.
Change from baseline in Standardized Asthma Quality of Life Questionnaire for 12 years and older (AQLQ(s)+12) total score at Week 28 | Baseline to Week 28
  Change from baseline in AQLQ(S)+12 as compared to placebo at Week 28. The AQLQ(S)+12 is a questionnaire that measures the health-related quality of life experienced by asthma subjects. The total score is defined as the average of all 32 questions in the AQLQ(S)+12 questionnaire. AQLQ(S)+12 is a 7-point scale questionnaire, ranging from 7 (no impairment) to 1 (severe impairment).
Change From Baseline in St George's Respiratory Questionnaire (SGRQ) Score at Week 28 | Baseline to Week 28
  Change from baseline in SGRQ as compared to placebo at Week 28. The questionnaire is divided into 2 parts: part 1 consists of 8 items pertaining to the severity of respiratory symptoms in the preceding 4 weeks; part 2 consists of 42 items related to the daily activity and psychosocial impacts of the individual's respiratory condition. The total score indicates the impact of disease on overall health status. This total score is expressed as a percentage of overall impairment, in which 100 represents the worst possible health status and 0 indicates the best possible health status.
Change from baseline in fractional exhaled nitric oxide (FeNO) at Week 28 | Baseline to Week 28
  Change from baseline in fractional exhaled nitric oxide (FeNO) at Week 28.
Change from baseline in peripheral blood eosinophils at Week 28 | Baseline to Week 28
  Change from baseline in blood eosinophil counts at Week 28.
Change from baseline in total serum immunoglobulin E (IgE) at Week 28 | Baseline to Week 28
  Change from baseline in total serum IgE at Week 28.
PK: Serum trough concentrations at Week 0, 12 and 28 | Baseline, Week 12 and Week 28
  Pharmacokinetics samples are collected at baseline and at Week 12 prior to study intervention administration, and at Week 28 (End of Treatment visit).
Immunogenicity: Incidence of anti-drug antibodies (ADA) at Week 0, 12, 28, and 40 | Baseline to Week 40
  Immunogenicity samples are collected at baseline and at Week 12 prior to study intervention administration, at Week 28 (End of Treatment visit) and at Week 40 (Follow-up visit). Persistently positive is defined as positive at >=2 post baseline assessments (with >=16 weeks between the first and the last positive) or positive at last post baseline assessment. Transiently positive is defined as having at least one post baseline ADA positive assessment and not fulfilling the conditions of persistently positive. Treatment boosted ADA defined as baseline positive ADA that was boosted to a 4 fold or higher level following treatment. Treatment emergent ADA defined as sum of treatment induced ADA and treatment boosted ADA.

CONTACTS AND LOCATIONS:
Locations (53):
- United States (9):
  - Research Site, Newport Beach, California
  - Research Site, Denver, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Hialeah, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Lincoln, Nebraska
  - Research Site, The Bronx, New York
  - Research Site, El Paso, Texas
  - Research Site, Kingwood, Texas
- Brazil (7):
  - Research Site, Botucatu
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São Bernardo do Campo
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Canada (2):
  - Research Site, Ajax, Ontario
  - Research Site, Québec, Quebec
- Chile (2):
  - Research Site, Curicó
  - Research Site, Santiago
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jindřichův Hradec
  - Research Site, Moravský Krumlov
  - Research Site, Olomouc
  - Research Site, Ostrava
- India (3):
  - Research Site, Ajmer
  - Research Site, Kanpur
  - Research Site, Vadodara
- Mexico (5):
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Monterrey
  - Research Site, San Luis Potosí City
  - Research Site, Veracruz
- Research Site, Lima, Peru
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Bychawa
  - Research Site, Bydgoszcz
  - Research Site, Chęciny
  - Research Site, Grudziądz
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Sosnowiec
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Suwon
- Thailand (3):
  - Research Site, Bang Kra So
  - Research Site, Bangkok
  - Research Site, Hat Yai
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluatedas per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes,indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level datain an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Call center number: 866-914-6996 Email address: az-asthmatrials@careboxhealth.com — https://asthmatrials.com/en-US